CLINICAL TRIAL: NCT06503627
Title: Incidence of Caesarean Scar Defect in Cases of Cesarean Section With and Without Bladder Flap Dissection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CS niche avoidance
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2023-07

CONDITIONS: CS Scar Defect(Niche) How to Avoid
Keywords: CSD-NICHE-avoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: closed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dissection of bladder flap for CS (Active Comparator)
  Interventions: Procedure: bladder flap dissection
- no dissection of bladder flap for CS (No Intervention)

INTERVENTIONS:
Procedure: bladder flap dissection — bladder flap dissection during caesarean section
  Arms: dissection of bladder flap for CS

SUMMARY:
Anatomically Uterine niche is an iatrogenic pouch-like defect at the site of previous caesarean scar due to defective tissue healing. Radiologically niche should be defined as an indentation at the site of the CS scar with a depth of at least 2 mm. A niche can be subclassified in: (1) simple niche; (2) simple niche with one branch; (3) complex niche (with more than one branch). (1-3) Uterine niche occurs in up to 70% women with previous cesarean of whom 30% are symptomatic. Reported prevalence varies: 24-70% with transvaginal sonography (TVS) and 56-84% with gel/saline instillation sonohysterography (SHG).This may be an underestimation because many women are asymptomatic and also because clinicians may not recognize niche as a cause of symptoms due to unawareness. Prevalence of 45.6% was reported in a prospective observational study (n = 371) where sonohysterography was done six months post-cesarean. Prevalence increases with increasing number of previous cesareans. (1-5) Potential Risk Factors Niche forms due to poor healing of cesarean scar. Risk factors are: (5-8)

1. Factors Affecting Lower Uterine Segment:

   Cervical dilatation of > 5 cm, > 5 h duration of labour and advanced fetal station predispose to large niche due to thinner or less vascularized myometrium resulting in inadequate healing(5,6)
2. Level of Uterine Incision Lower uterine incision towards the cervix results in poor healing, as mucus secreted by cervical glands interferes with myometrial approximation. Mucus accumulation gradually increases the niche size also (5,7) Cesarean section done in advanced labour after cervical effacement and also creation of uterovesical fold of peritoneum influence the level of uterine incision.
3. Uterine Closure Techniques Single-layer, decidua sparing closure technique predisposes to incomplete closure, compared to single full-thickness closure. A strong myometrial scar with proper anatomical approximation without tissue strangulation minimizes risk of niches (1,8) If muscular edges are thick, they are best approximated by including deeper part in the first layer and the remaining superficial cut edges in the second layer.

   Non-perpendicular sutures leading to an irregular myometrial closure, locking sutures or very tight second layer leading to ischemic necrosis result in poorly healed scar predisposing to niche formation.

   Thus, double-layer uterine closure using non-locking sutures is the optimal closure technique that results in thicker residual myometrium and hence potentially lower risk of niches.

   Suboptimal surgical techniques: Inadequate haemostasis, tissue ischemia, devascularization and excessive tissue manipulation contribute to poor scar healing and adhesions, consequently forming niche.
4. Adhesions Adhesion formation with abdominal wall pulls the uterine scar towards abdominal wall, exerting counteracting force opposite to the direction of retracting uterine scar tissue and causing impaired wound healing. This mechanism is encountered in non closure of peritoneum and creation of bladder flap that is not sutured. (7)
5. Retroflexed Uterus Effect of gravity on uterine corpus also increases counteracting forces. Large niches are mostly found with retroflexed uterus. (6,7)
6. Patient Factors Genetic predisposition contributes to impaired healing, inflammation, or adhesion formation, post-operative infection. (7) Gestational diabetes (odds ratio, 1.73), previous caesarean (OR, 3.14) and advanced body mass index (OR, 1.06) are independent risk factors. Risk increases by 6% for every additional unit increase in body mass index. (8)

Diagnosis:

Niche can be visualized in non-pregnant state using TVS, SHG, 3-D ultrasound, magnetic resonance imaging or hysteroscopy. An anechoic space at least 2 mm deep in the myometrium at caesarean scar site clinches the diagnosis. Niche Size and Residual Myometrium thickness are measured.

Residual myometrial thickness (RMT) is the vertical distance between uterine serosa and apex of defect. Large niches are defined when RMT is < 50% of adjacent myometrium or ≤ 2.2 mm on TVS. Absent residual myometrium is termed a total defect. (9,10)

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients who will undergo cesarean section for the first time (primi section)

Exclusion Criteria:

* 1- Patient with excessive adhesion that necessitate bladder dissection 2- Previous uterine surgery e.g. myomectomy 3- Patient with comorbidities affecting wound healing e.g. diabetes, autoimmune diseases , immunosuppression 4- Patient in active labour with cervical dilatation > 5cm

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — pregnant female patient candidate for CS
Enrollment: 250 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
incidence of CS niche(CS defect) | 3 months
  ultrasound detection and symptoms for CS NICHE

SECONDARY OUTCOMES:
AUB (abnormal uterine bleeding) complaint by the patients | 6 months
  abnormal uterine bleeding in cases of cs niche

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 months

REFERENCES:
- [Background] Kulshrestha V, Agarwal N, Kachhawa G. Post-caesarean Niche (Isthmocele) in Uterine Scar: An Update. J Obstet Gynaecol India. 2020 Dec;70(6):440-446. doi: 10.1007/s13224-020-01370-0. Epub 2020 Sep 21. PMID 33417629
- [Background] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016

DOCUMENTS (2):
  • Study Protocol (2023-04-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT06503627/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT06503627/SAP_001.pdf